CLINICAL TRIAL: NCT07361107
Title: Evaluation of Circulating Immune Response After Histosonics in Colorectal Cancer (ECHO-CRC)
Acronym: ECHO CRC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-0632
Record Dates: First submitted 2025-12-10; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Colorectal (Colon or Rectal) Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm (Experimental): This is a single-center, non-randomized, open-label, single-arm pilot study investigating the systemic immune response to histotripsy in patients with colorectal cancer with liver metastasis. Histotripsy is an FDA-approved, non-invasive therapeutic modality for the treatment of liver tumors, including both primary and metastatic lesions. In this study, we aim to evaluate the kinetics of peripheral T-cell response following histotripsy of colorectal cancer liver metastases (CRCLM).
  Given the well-documented immune-tolerant tumor microenvironment of liver metastases and their role in systemic resistance to checkpoint inhibitors, we hypothesize that histotripsy-induced tumor disruption will lead to measurable alterations in peripheral T-cell clonal expansion and exhaustion markers. We will assess these changes via serial blood draws before and after histotripsy, with the goal of characterizing the systemic immune impact of local tumor ablation. Findings from this study may inform future
  Interventions: Procedure: Histotripsy

INTERVENTIONS:
Procedure: Histotripsy — This is a single-center, non-randomized, open-label, single-arm pilot study investigating the systemic immune response to histotripsy in patients with colorectal cancer with liver metastasis. Histotripsy is an FDA-approved, non-invasive therapeutic modality for the treatment of liver tumors, including both primary and metastatic lesions. In this study, we aim to evaluate the kinetics of peripheral T-cell response following histotripsy of colorectal cancer liver metastases (CRCLM).
  Given the well-documented immune-tolerant tumor microenvironment of liver metastases and their role in systemic resistance to checkpoint inhibitors, we hypothesize that histotripsy-induced tumor disruption will lead to measurable alterations in peripheral T-cell clonal expansion and exhaustion markers. We will assess these changes via serial blood draws before and after histotripsy, with the goal of characterizing the systemic immune impact of local tumor ablation. Findings from this study may inform future

SUMMARY:
This is a single-center, non-randomized, open-label, single-arm pilot study investigating the systemic immune response to histotripsy in patients with colorectal cancer with liver metastasis. Histotripsy is an FDA-approved, non-invasive therapeutic modality for the treatment of liver tumors, including both primary and metastatic lesions. In this study, investigators aim to evaluate the kinetics of peripheral T-cell response following histotripsy of colorectal cancer liver metastases (CRCLM). Given the well-documented immune-tolerant tumor microenvironment of liver metastases and their role in systemic resistance to checkpoint inhibitors, investigators hypothesize that histotripsy-induced tumor disruption will lead to measurable alterations in peripheral T-cell clonal expansion and exhaustion markers. Investigators will assess these changes via serial blood draws before and after histotripsy, with the goal of characterizing the systemic immune impact of local tumor ablation. Findings from this study may inform future combination strategies integrating histotripsy with immunotherapy to enhance treatment response in microsatellite-stable CRC

DETAILED DESCRIPTION:
This is a single-center, non-randomized, open-label, single-arm pilot study investigating the systemic immune response to histotripsy in patients with colorectal cancer with liver metastasis. Histotripsy is an FDA-approved, non-invasive therapeutic modality for the treatment of liver tumors, including both primary and metastatic lesions. In this study, investigators aim to evaluate the kinetics of peripheral T-cell response following histotripsy of colorectal cancer liver metastases (CRCLM). Given the well-documented immune-tolerant tumor microenvironment of liver metastases and their role in systemic resistance to checkpoint inhibitors, investigators hypothesize that histotripsy-induced tumor disruption will lead to measurable alterations in peripheral T-cell clonal expansion and exhaustion markers. Investigators will assess these changes via serial blood draws before and after histotripsy, with the goal of characterizing the systemic immune impact of local tumor ablation. Findings from this study may inform future combination strategies integrating histotripsy with immunotherapy to enhance treatment response in microsatellite-stable CRC

ELIGIBILITY:
Inclusion Criteria:

* Gender: Both male and female patients will be eligible for enrollment.

  * Age at least 18 years.
  * Histologic (biopsy-proven) confirmation of metastatic microsatellite stable colorectal cancer with at least one radiographically evident hepatic metastasis.
  * Planned treatment with standard-of-care histotripsy.
  * Radiographic confirmation of hepatic metastases with computed tomography (CT) or magnetic resonance imaging (MRI), with CT preferred. Imaging must be performed within 60 days of the date of consent.
  * Adequate organ and marrow function as defined below:

    1. Absolute neutrophil count: ≥ 1,000/mcL
    2. Platelets: ≥ 100,000/mcL
    3. Total bilirubin ≤ 3x the upper limit of normal (ULN). This may be up to 5x ULN if Gilbert's syndrome is documented.
    4. AST and ALT ≤ 8x institutional ULN.
    5. Serum creatinine ≤ 2x ULN unless on dialysis.
  * Eastern Cooperative Oncology Group (ECOG) performance status 0 to 3.
  * Estimated life expectancy of at least 90 days as determined by the treating physician.
  * Demographic group: There are no restrictions based on race or ethnicity. Efforts will be made to ensure a representative patient population reflecting the diversity of individuals affected by CRCLM.
  * Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Major surgical procedure or significant traumatic injury within 14 days prior to histotripsy.

  * Therapy with an investigational drug within 14 days prior to histotripsy.
  * Clinically significant cardiovascular or cerebrovascular disease, including:

    * Myocardial infarction within 3 months prior to enrollment.
    * Unstable angina.
    * Congestive heart failure (New York Heart Association Classification Class > II).

      v. 3.0 22July2025 9
    * Serious cardiac arrhythmia (controlled atrial fibrillation or definitively treated arrhythmias via ablation are not considered exclusion criteria).
    * Cerebrovascular stroke with deficit within 3 months prior to enrollment.
  * Active infection requiring systemic therapy within 14 days prior to histotripsy, unless deemed to be a chronic disease state by the study PI.
  * Active pregnancy.
  * Patients with active infections, autoimmune diseases requiring systemic immunosuppression, or other uncontrolled comorbidities that could interfere with study participation will be excluded.
  * Severe cancer-associated cachexia that may interfere with systemic immune response, as assessed by the treating physician.
  * Any ongoing medical illness or injury that would significantly impact tolerability of therapy, including but not limited to:

    * Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture.
    * Clinical signs or symptoms of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding.
    * Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates histotripsy, may affect the interpretation of study results, or may render the patient at high risk for treatment complications.
  * Anyone that is unable to consent due to cognitive, psychological or other reasons that impact their capacity.
  * Deemed to be inappropriate for enrollment by the study PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2027-09-27 (Estimated); Study Completion 2027-09-27 (Estimated)

PRIMARY OUTCOMES:
Measure of System Immune Modulation via T-cells | 2 years
  To evaluate whether histotripsy of CRCLM induces systemic immune modulation, as measured by changes in peripheral T-cell clonal expansion and markers of T-cell exhaustion.
  Change in peripheral T-cell clonal expansion measured in the week prior to histotripsy, directly after histotripsy, and at 14, 28, and 90 days following histotripsy.
  Change in markers of T-cell exhaustion measured in the week prior to histotripsy, directly after histotripsy, and at 14, 28, and 90 days following histotripsy.

SECONDARY OUTCOMES:
Assess the Kinetics of Peripheral Immune Cell Response via T-cells | 2 years
  Change in the kinetics of T-cell clonal expansion measured at the week prior to histotripsy, directly after histotripsy, and at 14, 28, and 90 days following histotripsy via blood samples will be analyzed using statistical analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Zuckerberg Cancer Center, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided